CLINICAL TRIAL: NCT00612742
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study of the Long-Term Safety and Efficacy of LibiGel® for the Treatment of Hypoactive Sexual Desire Disorder in Postmenopausal Women
Brief Title: Safety and Efficacy of LibiGel® for Treatment of Hypoactive Sexual Desire Disorder in Postmenopausal Women
Acronym: BLOOM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioSante Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TESTW007
Record Dates: First submitted 2008-01-23; First posted 2008-02-12 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: Cardiovascular event; Breast Cancer; Testosterone; Menopause; Hypoactive Sexual Desire Disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Breast Neoplasms | interventions — Testosterone Propionate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- testosterone gel (Experimental): 1% testosterone transdermal gel
  Interventions: Drug: testosterone gel
- placebo gel (Placebo Comparator): placebo transdermal gel
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: testosterone gel — once daily transdermal testosterone gel, 300 mcg
  Other Names: LibiGel
  Arms: testosterone gel
Drug: placebo gel — once daily transdermal placebo gel
  Arms: placebo gel

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, adaptive design, multi-center study of the long-term cardiovascular and breast safety of LibiGel in the treatment of HSDD in postmenopausal women with at least two points of cardiovascular risk and clinical diagnosis of Hypoactive Sexual Desire Disorder (HSDD).

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal female subjects

* at least 50 years of age
* with at least two points of cardiovascular risk
* with a clinical diagnosis of HSDD.

Exclusion Criteria:

Subjects must not

* require treatment with anti-androgens, high-dose oral or injectable corticosteroids, tamoxifen or other selective estrogen receptor modulators,
* have used androgen therapy within 2 months of randomization,
* have a history of estrogen-dependent neoplasia or any gynecologic cancer,
* have a history of cancer of any kind in the past 10 years prior to randomization,
* have a history of malignant melanoma or a history of invasive cancer at any time,
* have a screening mammogram with any finding that requires follow up within 6 months of randomization,
* have a history of myocardial infarction, coronary revascularization or stroke within 12 months of randomization,
* have any medical condition associated with predicted survival of less than 3 years in the judgment of the Investigator.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3656 (Actual)
Dates: Start 2008-01; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The rate of adjudicated, predefined cardiovascular events in LibiGel-treated subjects compared to that of placebo-treated subjects. | 2011 primary outcome analysis for NDA submission

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Snabes, MD, PhD, Study Director — BioSante Pharmaceuticals, Inc.
Locations (149):
- United States (141):
  - BioSante Site #215, Birmingham, Alabama
  - BioSante Site 185, Birmingham, Alabama
  - BioSante Site 095, Hoover, Alabama
  - BioSante Site #014, Huntsville, Alabama
  - BioSante Site 196, Huntsville, Alabama
  - BioSante Site 146, Mobile, Alabama
  - BioSante Site 171, Chandler, Arizona
  - BioSante Site 145, Glendale, Arizona
  - BioSante Site 027, Glendale, Arizona
  - BioSante Site 121, Phoenix, Arizona
  - BioSante Site 137, Tucson, Arizona
  - BioSante Site 040, Tucson, Arizona
  - BioSante Site 052, Hot Springs, Arkansas
  - BioSante Site 100, Jonesboro, Arkansas
  - BioSante Site #060, Little Rock, Arkansas
  - BioSante Site 155, Little Rock, Arkansas
  - BioSante Site 011, Los Angeles, California
  - BioSante Site 094, Palm Springs, California
  - BioSante Site 043, Roseville, California
  - BioSante Site 162, Sacramento, California
  - BioSante Site 025, Sacramento, California
  - BioSante Site 112, San Diego, California
  - BioSante Site 008, San Diego, California
  - BioSante Site #070, San Diego, California
  - BioSante Site 205, San Diego, California
  - BioSante Site #192, San Diego, California
  - BioSante Site 159, Walnut Creek, California
  - BioSante Site 007, Denver, Colorado
  - BioSante Site 216, Denver, Colorado
  - BioSante Site 026, Lakewood, Colorado
  - BioSante Site 166, Farmington, Connecticut
  - BioSante Site 103, Hartford, Connecticut
  - BioSante Site 132, New Britain, Connecticut
  - BioSante Site 151, New London, Connecticut
  - BioSante Site 036, Ridgefield, Connecticut
  - BioSante Site 013, Washington D.C., District of Columbia
  - BioSante Site 118, Aventura, Florida
  - BioSante Site 139, Crystal River, Florida
  - BioSante Site 143, Jacksonville, Florida
  - BioSante Site 180, Melbourne, Florida
  - BioSante Site 024, Miami, Florida
  - BioSante Site #219, Pinellas Park, Florida
  - BioSante Site 041, St. Petersburg, Florida
  - BioSante Site 152, Tampa, Florida
  - BioSante Site 009, West Palm Beach, Florida
  - BioSante Site 115, Atlanta, Georgia
  - BioSante Site 017, Meridian, Idaho
  - BioSante Site 189, Addison, Illinois
  - BioSante Site 156, Champaign, Illinois
  - BioSante Site 045, Chicago, Illinois
  - BioSante Site 149, Chicago, Illinois
  - BioSante Site 133, Chicago, Illinois
  - BioSante Site 167, Newburgh, Indiana
  - BioSante Site 022, South Bend, Indiana
  - BioSante Site 163, Overland Park, Kansas
  - BioSante Site #214, Lexington, Kentucky
  - Biosante Site #136, Lexington, Kentucky
  - BioSante Site 005, Shreveport, Louisiana
  - BioSante Site 004, Baltimore, Maryland
  - BioSante Site 195, Greenbelt, Maryland
  - BioSante Site 066, Rockville, Maryland
  - BioSante Site #206, Fall River, Massachusetts
  - BioSante Site 035, Ann Arbor, Michigan
  - BioSante Site 124, Bingham Farms, Michigan
  - BioSante Site 044, Detroit, Michigan
  - BioSante Site 047, Grand Rapids, Michigan
  - BioSante Site 105, Paw Paw, Michigan
  - BioSante Site 033, Saginaw, Michigan
  - BioSante Site 031, Saint Clair Shores, Michigan
  - BioSante Site #208, Edina, Minnesota
  - BioSante Site 198, Saint Paul, Minnesota
  - BioSante Site 081, Olive Branch, Mississippi
  - BioSante Site 104, St Louis, Missouri
  - BioSante Site 127, Billings, Montana
  - BioSante Site 051, Missoula, Montana
  - BioSante Site 006, Lincoln, Nebraska
  - BioSante Site 018, Las Vegas, Nevada
  - BioSante Site #217, Las Vegas, Nevada
  - BioSante Site 125, Lawrenceville, New Jersey
  - BioSante Site 179, Albuquerque, New Mexico
  - BioSante Site 019, New York, New York
  - BioSante Site 015, Poughkeepsie, New York
  - BioSante Site 161, Purchase, New York
  - BioSante Site 079, Charlotte, North Carolina
  - BioSante Site 072, Hickory, North Carolina
  - BioSante Site 107, Raleigh, North Carolina
  - BioSante Site 034, Winston-Salem, North Carolina
  - BioSante Site 058, Winston-Salem, North Carolina
  - BioSante Site 061, Winston-Salem, North Carolina
  - BioSante Site 131, Winston-Salem, North Carolina
  - BioSante Site 056, Fargo, North Dakota
  - BioSante Site 071, Minot, North Dakota
  - BioSante Site #210, Akron, Ohio
  - BioSante Site #130, Beachwood, Ohio
  - BioSante Site #212, Cincinnati, Ohio
  - BioSante Site 101, Cleveland, Ohio
  - BioSante Site #213, Columbus, Ohio
  - BioSante Site 160, Englewood, Ohio
  - BioSante Site 153, Gallipolis, Ohio
  - BioSante Site 116, Mayfield Heights, Ohio
  - BioSante Site 138, West Chester, Ohio
  - BioSante Site 129, Tulsa, Oklahoma
  - BioSante Site #050, Eugene, Oregon
  - BioSante Site #106, Eugene, Oregon
  - BioSante Site 126, Medford, Oregon
  - BioSante Site #203, Portland, Oregon
  - BioSante Site 165, Jenkintown, Pennsylvania
  - BioSante Site 142, Pittsburgh, Pennsylvania
  - BioSante Site 099, Sellersville, Pennsylvania
  - BioSante Site 074, West Reading, Pennsylvania
  - BioSante Site 075, Warwick, Rhode Island
  - BioSante Site 117, Anderson, South Carolina
  - BioSante Site 089, Columbia, South Carolina
  - BioSante Site #209, Greer, South Carolina
  - BioSante Site 097, Hilton Head Island, South Carolina
  - BioSante Site 038, Mt. Pleasant, South Carolina
  - BioSante Site 093, Bristol, Tennessee
  - BioSante Site 069, Chattanooga, Tennessee
  - BioSante Site 002, Germantown, Tennessee
  - BioSante Site 078, Memphis, Tennessee
  - BioSante Site 042, Nashville, Tennessee
  - BioSante Site 048, Austin, Texas
  - BioSante Site 073, Corpus Christi, Texas
  - BioSante Site #220, Dallas, Texas
  - BioSante Site 147, Dallas, Texas
  - BioSante Site 039, Houston, Texas
  - BioSante Site 122, Houston, Texas
  - BioSante Site 154, Hurst, Texas
  - BioSante Site #211, San Antonio, Texas
  - BioSante Site 084, San Antonio, Texas
  - BioSante Site #218, Murray, Utah
  - BioSante Site 102, Salt Lake City, Utah
  - BioSante Site 168, Sandy City, Utah
  - BioSante Site 096, Williston, Vermont
  - BioSante Site 003, Charlottesville, Virginia
  - BioSante Site 086, Norfolk, Virginia
  - BioSante Site 053, Richmond, Virginia
  - BioSante Site 090, Virginia Beach, Virginia
  - BioSante Site #083, Mountlake Terrace, Washington
  - BioSante Site 128, Seattle, Washington
  - BioSante Site #158, Milwaukee, Wisconsin
- Canada (8):
  - BioSante Site #175, Vancouver, British Columbia
  - BioSante Site #164, Winnipeg, Manitoba
  - BioSante Site 190, Hamilton, Ontario
  - BioSante Site #088, Newmarket, Ontario
  - BioSante Site 088, Newmarket, Ontario
  - BioSante Site 188, Sarnia, Ontario
  - BioSante Site 054, Windsor, Ontario
  - BioSante Site 109, Québec, Quebec

REFERENCES:
- [Derived] White WB, Grady D, Giudice LC, Berry SM, Zborowski J, Snabes MC. A cardiovascular safety study of LibiGel (testosterone gel) in postmenopausal women with elevated cardiovascular risk and hypoactive sexual desire disorder. Am Heart J. 2012 Jan;163(1):27-32. doi: 10.1016/j.ahj.2011.09.021. Epub 2011 Nov 21. PMID 22172433
- See also: www.Bloom study.com Click here for more information about this study: Safety and Efficacy of LibiGel® for Treatment of Hypoactive Sexual Desire Disorder in Postmenopausal Women — http://www.bloomstudy.com